CLINICAL TRIAL: NCT00167505
Title: SIP 4-04 Evaluation of Abstinence-Only and Abstinence-Plus Program to Prevent HIV, STD, and Pregnancy Among Middle School Students
Brief Title: All About Youth: Evaluation of Sexual Risk Avoidance and Risk Reduction Programs for Middle School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Christine Markham, PhD, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U48DP000057 (NIH); NCT00167505; NCT00207545 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Sexually Transmitted Diseases; Pregnancy; HIV Infections
Keywords: adolescents; sexual health; HIV; STD; pregnancy prevention; abstinence education; HIV Seronegativity; human immunodeficiency virus
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risk Avoidance (Experimental): The risk avoidance intervention is a Title V compliant curriculum emphasizing abstinence until marriage and strong character development. The curriculum includes both classroom and CD-ROM based lessons delivered in the 7th and 8th grade. Lessons include topics such as puberty, reproduction, healthy relationships, consequences of sex, and refusal skills.
  Interventions: Behavioral: Risk Avoidance Intervention
- Risk Reduction (Experimental): The risk reduction intervention is a curriculum providing skills for abstinence and condom and other contraceptive use. The curriculum includes both classroom and CD-ROM based lessons delivered in the 7th and 8th grade. Lessons include topics such as puberty, reproduction, healthy relationships, consequences of sex, and refusal skills.
  Interventions: Behavioral: Risk Reduction Intervention

INTERVENTIONS:
Behavioral: Risk Avoidance Intervention — The risk avoidance intervention is a Title V compliant curriculum emphasizing abstinence until marriage and strong character development. The curriculum includes 12 classroom and CD-ROM based lessons delivered in the 7th and 8th grade. Lessons include topics such as puberty, reproduction, healthy relationships, consequences of sex, and refusal skills.
  Arms: Risk Avoidance
Behavioral: Risk Reduction Intervention — The risk reduction intervention is a curriculum providing skills for abstinence and condom and other contraceptive use. The curriculum includes 12 classroom and CD-ROM based lessons delivered in the 7th and 8th grade. Lessons include topics such as puberty, reproduction, healthy relationships, consequences of sex, and refusal skills.
  Arms: Risk Reduction

SUMMARY:
This study will evaluate the efficacy of two curricula relative to standard care. The first is a sexual risk avoidance curriculum for middle school students that included abstinence until marriage and complies with Title V Section 510 A-H abstinence education requirements. The second is a sexual risk reduction curriculum for middle school students that included abstinence and condom/contraceptive information and skills. Each intervention consists of an age-appropriate classroom curriculum and a CD-ROM-based tailored intervention delivered in 7th and 8th grade. The overall goal of the study is to identify common elements of effective sexuality education curricula that will be of benefit to youth.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of a risk avoidance program for middle school students and a theoretically-comparable risk reduction program relative to standard care. The study design is a randomized controlled trial conducted in fifteen inner-city middle schools in Houston, Texas. Five schools were randomly assigned to a risk avoidance intervention, five to a risk reduction intervention, and five to a comparison (standard care) condition. Approximately, 1,800 7th grade students were recruited into the study and will be followed over a three-year period. Based on a formative study, a pilot study, and input from community groups and a national panel of experts, two comparable curricula were developed. The risk avoidance curriculum emphasizes sexual abstinence until marriage and includes the requirements for abstinence education as defined in Title V, Section 510. The risk reduction curriculum emphasizes abstinence and addresses condom and contraceptive use. The risk avoidance and risk reduction interventions each consist of an age-appropriate classroom curriculum and a CD-ROM-based tailored intervention delivered in 7th and 8th grade. Each intervention was delivered by trained facilitators. The effect of the interventions will be evaluated by assessing sexual risk-taking behaviors of participants in each intervention (proportion of students initiating sexual intercourse, proportion that are sexually active, number of times of unprotected sex, number of sexual partners) relative to the comparison group. Risk assessment data from students was collected by using an audio computer-assisted self-interview (ACASI) approach for the collection of baseline, 6-, 18-, and 24-month data. Parental permission and child assent were required prior to participation. In addition, we will conduct a 36-month follow-up survey and a one-time urine-based test for chlamydia, gonorrhea, and trichomonas which will provide additional longitudinal data to assess the impact of each curriculum, relative to standard care.

ELIGIBILITY:
Inclusion Criteria:

* 7th graders attending regular classes in Houston Independent School District

Exclusion Criteria:

* No students will be excluded based on race/ethnicity, age, or gender
* Students will be informed that the surveys and intervention materials will only be available in English and will be asked to consider their comfort level with participating in the study.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1742 (Actual)
Dates: Start 2006-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
delay onset of sex | baseline, 6,18, 24, and 36 month follow-up

SECONDARY OUTCOMES:
knowledge | baseline, 6,18, 24, and 36 month follow-up
skills | baseline, 6, 18, 24, and 36 month follow-up
self-efficacy | baseline, 6, 18, 24, and 36 month follow-up
attitudes | baseline, 6, 18, 24, and 36 month follow-up
condom use | baseline, 6, 18, 24, and 36 month follow-up
alcohol/drug use | baseline, 6, 18, 24, and 36 month follow-up
number of sexual partners | baseline, 6, 18, 24, and 36 month follow-up
prevalence of chlamydia, gonorrhea, and trichomonas | 36-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christine Markham, PhD, Principal Investigator — University of Texas Houston School of Public Health
Locations (1):
- University of Texas Houston School of Public Health, Houston, Texas, United States